CLINICAL TRIAL: NCT04868786
Title: Population Pharmacokinetic and Pharmacodynamic Model-based Dosing Strategy of Mycophenolate Mofetil in Pediatric Hematopoietic Stem Cell Transplantation(HSCT) Patients
Brief Title: Pharmacokinetics and Pharmacodynamics of Mycophenolate Mofetil in Pediatric Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Institute of Food and Drug Safety Evaluation (Republic of Korea) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SNUCH-MIDD-MMF
Record Dates: First submitted 2021-03-28; First posted 2021-05-03 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mycophenolate Mofetil (Experimental)
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Administer 15-20mg/kg of mycophenolate mofetil twice daily. Blood sampling for pharmacokinetics(PK) of mycophenolate mofetil will be performed in all patients who have taken the investigational drug for at least 3 days.

SUMMARY:
This is an investigator-initiated clinical trial to analysis population pharmacokinetic characteristics and investigate appropriate pediatric dose of mycophenolate mofetil in pediatric hematopoietic stem cell transplantation patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had mycophenolate treatment at least 3 days for immunosuppressant after allogenic hematopoietic stem cell transplantation
* Patients age <18 years
* Written Study Informed consent and/or assent from the patient, parent, or guardian

Exclusion Criteria:

* Known hypersensitivity to mycophenolate mofetil or similar class of drug substance
* Patients in medically critical condition such as severe infection or unstable vital signs
* Any condition that would, in the Investigator's judgment, interfere with full participation in the study
* Patients with hypoxanthine-guanine phosphoribosyltransferase deficiency(HGPRT) such as Lesch-Nyhan or Kelley-Seegmiller syndrome)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics parameter of melphalan | pre dose, post 1 hour, post 2 hour, post 6 hour
  Analysis: Maximum plasma drug concentration (Cmax)
Pharmacokinetics parameter of melphalan | pre dose, post 1 hour, post 2 hour, post 6 hour
  Analysis: Time to reach maximum plasma concentration (tmax)
Pharmacokinetics parameter of melphalan | pre dose, post 1 hour, post 2 hour, post 6 hour
  Analysis: Area under the plasma concentration-time curve (AUC)
Pharmacokinetics parameter of melphalan | pre dose, post 1 hour, post 2 hour, post 6 hour
  Analysis: Apparent total clearance of the drug from plasma after oral administration (CL/F)
Pharmacokinetics parameter of melphalan | pre dose, post 1 hour, post 2 hour, post 6 hour
  Analysis: Apparent volume of distribution after non-intravenous administration (V/F)

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea